CLINICAL TRIAL: NCT04411407
Title: Patient-reported Outcome Measures Collected in DANBIO Via a From Home Web Application Versus a Touchscreen in the Outpatient Clinic Among Patients With Systemic Lupus Erythematosus: A Randomised, Crossover, Agreement Study
Brief Title: PROM Collected Via a WebApp Versus a Touch Screen Solution Among Patients With SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salome Kristensen (Other)
Responsible Party: Sponsor-Investigator, Salome Kristensen, Chief physician, PhD, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20200527
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: A randomised, within-participants, open, cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group WT (Other): PROM registration via the DANBIO WebApp and thereafter the outpatient touchscreen
  Interventions: Device: PROM registration via the DANBIO WebApp and the outpatient touchscreen in a randomised order
- Group TW (Other): PROM registration via the outpatient touchscreen and thereafter the DANBIO WebApp
  Interventions: Device: PROM registration via the DANBIO WebApp and the outpatient touchscreen in a randomised order

INTERVENTIONS:
Device: PROM registration via the DANBIO WebApp and the outpatient touchscreen in a randomised order — PROM registration via the DANBIO WebApp and the outpatient touchscreen in a randomised order

SUMMARY:
A randomised, within-participants cross-over design trial including 34 patients with systemic lupus erythematosus. The participants will be randomised to data registration of patient reported outcome measures (PROM) through the DANBIO webapp and thereafter via the outpatient touchscreen or vice versa.

DETAILED DESCRIPTION:
The aim of this trial is to evaluate whether electronic reporting of PROMs through the DANBIO web application (webapp) is comparable to the outpatient touchscreen among patients with SLE.

The trial is a randomised, crossover, agreement study where 34 patients with SLE from the Department of Rheumatology at Aalborg University Hospital will be included and randomised in ratio 1:1 to:

* Group 1: PROMs are reported through the DANBIO webapp; thereafter, the touchscreen.
* Group 2: PROMs are reported through the touchscreen; thereafter, the DANBIO webapp.

There will be a wash-out period of 1-2 day between the two registrations to minimise carryover bias.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed in DANBIO with SLE
* Experience with the PROM questionnaires in DANBIO (≥ 1 previous assessments)

Exclusion Criteria:

* Inability to provide informed consent or to comply with the study protocol
* Diagnosis of SLE of ≥ 12 months
* Does not have access to a device that can run the DANBIO webapp

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Systemic Lupus Activity Questionnaire global health | Day 1 (first data registration) and day 3 (second data registration)
  Evaluates global assessment of lupus activity using an NRS score from 0-10. Higher score Means worse outcome.

SECONDARY OUTCOMES:
Change in Health Assessment Questionnaire (HAQ) | Day 1 (first data registration) and day 3 (second data registration)
  Assess the patient's physical function from 0-3. Higher score Means worse outcome.
Visual Analogue Scale for Pain | Day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of pain on a scale from 0-100 within the last week.The left of the scale (0) signifies the absence of pain and the right end (100) maximum pain.
Visual Analogue Scale for fatigue | Day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of fatigue on a scale from 0-100 within the last week. The left of the scale (0) signifies the absence of fatigue and the right end (100) maximum fatigue.
Patient Global Visual Analogue Scale | Day 1 (first data registration) and day 3 (second data registration)
  The patient's global assessment of disease activity (arthritis severity) on a scale from 0-100 within the last week. The left of the scale (0) signifies the absence of arthritis activity and the right end (100) maximum arthritis activity.
Patient Acceptable Symptom State (PASS) | Day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of acceptable symptom state. Consist of one question answered with "yes" or "no". The question is: ''Take into account all the ways in which your arthritis has affected you in the past 48 hours. If you were to remain for the next few months as you are today, would it be acceptable to you?"
Anchoring question | Day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of change in arthritis activity since last visit from much worse to much better.
SLAQ flare score | Day 1 (first data registration) and day 3 (second data registration)
  Evaluates presence or severity of lupus flare on a transitional scale e.g. 0 (no worsening), 1 (mild worsening), 2 (moderate worsening) or 3 (severe worsening).
SLAQ symptom score | Day 1 (first data registration) and day 3 (second data registration)
  Evaluates the number of lupus specific symptoms present from 0-24. Higher score means worse outcome.
SLAQ total score | Day 1 (first data registration) and day 3 (second data registration)
  Evaluates severity of lupus disease activity by a weighted score of the 24 lupus specific symptoms, range 0-44. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kristensen, MD, PhD, Principal Investigator — Department of Rheumatology, Aalborg University Hospital
Locations (1):
- Department of Rheumatology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and the SAP will be published as supplementary information to the article. IPD from this trial that underlie results in a publication will be made available in clinicaltrials.gov after publication of the article.
Supporting Information: Study Protocol, SAP
Time Frame: Will be made available when the article is published
Access Criteria: Study protocol and the SAP will be published as supplementary information to the article. IPD from this trial that underlie results in a publication will be made available in clinicaltrials.gov after publication of the article.